CLINICAL TRIAL: NCT04540445
Title: Utility of Pupillary Metrics in Diagnosis and Management of Concussion in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: NeurOptics Inc. (Industry)
Responsible Party: Principal Investigator, Theodore Heyming, Principal Investigator, Children's Hospital of Orange County
Other Study IDs: 1909112
Record Dates: First submitted 2020-02-27; First posted 2020-09-07 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Brain Concussion; Reflex, Pupillary; Post-Concussion Syndrome; Brain Injuries, Traumatic
Keywords: pupillometry; concussion; traumatic brain injury; post-concussion syndrome
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Concussed Cohort: The concussed cohort will consist of children ages 5-17 diagnosed with a concussion within 72 hours following injury and recruited from a pediatric emergency department.
  Interventions: Other: Pupillary Assessment
- Healthy Matched Controls: The healthy matched control cohort consists of children 5-17, who are age and gender matched to concussed subjects who will be recruited from affiliated pediatric primary care and adolescent clinics.
  Interventions: Other: Pupillary Assessment

INTERVENTIONS:
Other: Pupillary Assessment — Pupillary assessment with handheld pupillometer
  Other Names: NeurOptics PLR-3000; NeurOptics NPi®-200

SUMMARY:
The purpose of this study is to gather information and compare the potential use of pupillometry to identify concussions and post concussive syndrome with standard age appropriate assessments. The study will compare concussed pediatric patients 5-17 years of age recruited from the emergency department within 72 hours following injury with age and gender matched non-concussed pediatric patients recruited from primary care clinics. Assessment of both concussed and non-concussed subjects will take place at the initial enrollment visit and will be repeated at 1-2 weeks for the concussed subjects and at 12-14 weeks for both groups.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is the leading cause of disability and death in children. In both pediatric and adult populations, concussion is the most prevalent type of TBI and can result in persistent post-concussive symptoms. Early recognition and treatment of concussion is critical to the prevention of long-term sequelae and has recently become a national public-health priority. Comprehensive assessment and diagnosis of concussion commonly includes the use of a multimodal approach using a graded symptoms checklist, neurocognitive testing, and balance assessment. An objective biomarker to definitively diagnose concussion would revolutionize its management-allowing for accurate and immediate determination of return to play/duty, decreasing unnecessary exposure to radiation, and reducing the overall cost of care. Considering the paucity of evidence regarding the use of pupillary light reflex in concussed children and the lack of a biomarker for concussion, further examination of the use of objective pupillary metrics in this population is warranted.

The purpose of this study is to gather information and compare the potential use of pupillometry to identify concussions and post concussive syndrome with standard age appropriate assessments. The proposed study design is prospective, longitudinal case-control consisting of two distinct cohorts: concussed participants and healthy control participants. All concussion management decisions will be determined independent of the study by the healthcare provider(s). Trained personnel performing follow-up assessments will use established clinical criteria to notify appropriate healthcare provider and/or study team member of any clinical concerns or unanticipated events.

The study will compare concussed pediatric patients 5-17 years of age recruited from the emergency department within 72 hours following injury with age and gender matched non-concussed pediatric patients recruited from affiliated primary care and adolescent clinics. Assessment of both concussed and non-concussed subjects will take place at the initial enrollment visit and will be repeated at 1-2 weeks for the concussed subjects and at 12-14 weeks for both groups. Age appropriate assessment will include the Post-Concussion Symptom Inventory (PCSI), Post-Concussion Symptom Scale (PCSS), pupillometry, Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT), and Balance Error Scoring System (BESS).

The primary objectives are to examine the acute (<72 hours), subacute (1-2 week), and long-term (12-14 weeks post-injury) longitudinal association among pupillary metrics, standardized neurocognitive tests, and objective balance assessment in pediatric patients with concussion versus controls. The secondary objectives are to evaluate the effectiveness of pupillometer data as an objective biomarker to aid in the identification of concussion and post-concussive syndrome in children. Results will generate new knowledge regarding the clinical utility of pupillometers in this patient population. We will explore the period that best differentiates concussion and controls.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 5 to < 18 years of age
2. Patients presenting to Pediatric Emergency Department with a concussion within 72 hours following injury. Concussion will be defined as the presence of the following criteria: Post injury patient reported symptoms on an age-appropriate graded-symptom checklist that meets the borderline to extremely high threshold (sex and age adjusted)
3. Age and gender matched healthy controls recruited and evaluated through Primary Care (Orange Ambulatory) and Adolescent Clinics

Exclusion Criteria:

1. Lower extremity deficiency or injury
2. History of cognitive deficiencies
3. History of ≥ 3 prior concussions
4. History of attention deficit disorder
5. Previously diagnosed concussion within the past year
6. History of intracranial disease
7. History of unresolved strabismus, diplopia, amblyopia
8. History of unresolved cranial nerve III, IV or VI palsy
9. History of unresolved macular edema, retinal degeneration, extensive cataract, or ocular globe disruption
10. History of unresolved extensive corneal surgery or scarring
11. Lack of two functional eyes
12. Unresolved oculo-motor dysfunctions
13. Obvious intoxication or impairment that limits ability to participate
14. Imaging abnormality (i.e. fracture or bleed)
15. Color blindness OR failing the Ishihara screening for color blindness
16. Unable to come in for follow-up visits
17. In addition to the above exclusion criteria, healthy control participants will be excluded if they have a history of chronic disease.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will consist of concussed patients ages 5-17 presenting at a pediatric emergency department within 72 hours following concussion and healthy controls that are age and gender matched to concussed subjects recruited from affiliated primary care and adolescent clinics.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The association between NPi®-200 pupillometer measurements (including variables such as size, latency, constriction velocity, dilation velocity, etc.) and concussed/control status over time. | For concussed subjects: the first measurement will be within 72 hours of sustaining injury, then repeated at 1-2 weeks and at 12-14 weeks post injury. For control subjects: the first measurement will be at enrollment and repeated at 12-14 weeks.
  NPi®-200 pupillometer is a hand-held portable infrared device which provides quantitative pupillary measurements by taking 30 pictures per second of the pupil's response to light stimulus for a duration of 3 seconds. A patient's pupil measurement (including variables such as size, latency, constriction velocity, dilation velocity, etc.) is compared against a normative model of pupil reaction to light and automatically graded by the Neurological Pupil Index (NPi™) on a scale of 0 to 5. Pupillary measurements will be obtained for the right and left eye.
The association between the NeurOptics PLR-3000 pupillometer measurements (including variables such as size, latency, constriction velocity, dilation velocity, etc.) and concussed/control status over time. | For concussed subjects: the first measurement will be within 72 hours of sustaining injury, then repeated at 1-2 weeks and at 12-14 weeks post injury. For control subjects: the first measurement will be at enrollment and repeated at 12-14 weeks.
  The NeurOptics PLR-3000 pupillometer is a hand-held portable infrared device which provides quantitative pupillary measurements by taking 30 pictures per second of the pupil's response to light stimulus for a duration of 6 seconds. Pupillary data, such as constriction velocity, latency, pupil size before and after the reflex, dilation velocity, time to reach 75% of initial resting diameter after constriction (T75) are calculated automatically at the end of each measurement. Pupillary measurements will be obtained for the right and left eye.
The association between the Post-Concussion Symptom Inventory (PCSI) & Post-Concussion Symptom Scale (PCSS) and concussed/control status over time. | For concussed subjects: the first measurement will be within 72 hours of sustaining injury, then repeated at 1-2 weeks and at 12-14 weeks post injury. For control subjects: the first measurement will be at enrollment and repeated at 12-14 weeks.
  PCSI assesses post-concussion symptoms based on patient and parent/teacher report. This inventory focuses on four areas that may be affected after concussion: cognitive, emotional, physical, and sleep. There are age-specific forms available for children between 5-7 years old, 8-12 years old, and 13-18 years old. This tool has been found to have moderate to high (0.62 to 0.84) inter-rater reliability for child reports and internal consistency across the three reports.
  PCSS is also a self-reported assessment of post-concussion symptoms. This report, which is part of the widely used Sport Concussion Assessment Tool (SCAT) Versions 3 and 5 and Immediate Post-Concussion Assessment and Cognitive Test (ImPACT), quantifies symptom severity (rank 22 different possible post-concussion symptoms on 7 point Likert scale). Similar to the PCSI, the PCSS includes symptoms from four areas: cognitive, emotional, physical, and sleep.
The association between the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT®) & ImPACT® Pediatric assessment and concussed/control status over time. | For concussed subjects: the first measurement will be within 72 hours of sustaining injury, then repeated at 1-2 weeks and at 12-14 weeks post injury. For control subjects: the first measurement will be at enrollment and repeated at 12-14 weeks.
  ImPACT® and ImPACT® Pediatric will both be used in this study. ImPACT® is a computerized data collection and neuropsychological testing tool commonly used for baseline and post-injury testing in athletes (12-59 years of age) at risk for sports-related concussion. Subjects participate in neuropsychological tests which assess attention, verbal memory, visual memory, visual processing speed, and reaction times. ImPACT® will be used to evaluate study patients ≥12 years old. ImPACT® Pediatric is an examiner-administered iOS-based battery of neuropsychological tests designed to measure neurocognitive functioning in children ages 5-11. ImPACT® Pediatric is administered on an iPad and is a neurocognitive test for management of pediatric concussions. ImPACT® Pediatric will be used to evaluate patients < 12 years old. Outcome variables will be obtained from ImPACT® and include data to evaluate: verbal memory, visual memory, visual processing speed, and reaction time.
The association between the Balance Error Scoring System (BESS) scores and concussed/control status over time. | For concussed subjects: the first measurement will be within 72 hours of sustaining injury, then repeated at 1-2 weeks and at 12-14 weeks post injury. For control subjects: the first measurement will be at enrollment and repeated at 12-14 weeks.
  The Balance Error Scoring System (BESS) provides an objective score for a patient's postural stability. The patient is instructed to stand in three different stances, first on a solid surface and then a foam surface, for 20 seconds each. The examiner records the number of errors, as predefined by the scoring system, during each stance. The maximum score is 60 and a higher score correlates with worsening postural stability. This test has demonstrated good test-rest reliability (0.87-0.97 intraclass correlations), low to moderate sensitivity (0.34 to 0.64), and high specificity (0.91). Sensitivity is increased when this test is used in conjunction with a graded symptom checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Heyming, MD, Principal Investigator — CHOC Children's Hospital of Orange County
Locations (1):
- CHOC Children's, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available as data may be proprietary in nature.

REFERENCES:
- [Background] Schutzman SA, Greenes DS. Pediatric minor head trauma. Ann Emerg Med. 2001 Jan;37(1):65-74. doi: 10.1067/mem.2001.109440. PMID 11145776
- [Background] Bazarian JJ, McClung J, Shah MN, Cheng YT, Flesher W, Kraus J. Mild traumatic brain injury in the United States, 1998--2000. Brain Inj. 2005 Feb;19(2):85-91. doi: 10.1080/02699050410001720158. PMID 15841752
- [Background] Wortzel HS, Granacher RP Jr. Mild Traumatic Brain Injury Update: Forensic Neuropsychiatric Implications. J Am Acad Psychiatry Law. 2015 Dec;43(4):499-505. PMID 26668228
- [Background] Zaloshnja E, Miller T, Langlois JA, Selassie AW. Prevalence of long-term disability from traumatic brain injury in the civilian population of the United States, 2005. J Head Trauma Rehabil. 2008 Nov-Dec;23(6):394-400. doi: 10.1097/01.HTR.0000341435.52004.ac. PMID 19033832
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] Papa L. Potential Blood-based Biomarkers for Concussion. Sports Med Arthrosc Rev. 2016 Sep;24(3):108-15. doi: 10.1097/JSA.0000000000000117. PMID 27482776
- [Background] Burke MJ, Fralick M, Nejatbakhsh N, Tartaglia MC, Tator CH. In search of evidence-based treatment for concussion: characteristics of current clinical trials. Brain Inj. 2015;29(3):300-5. doi: 10.3109/02699052.2014.974673. Epub 2014 Nov 10. PMID 25383510
- [Background] Bin Zahid A, Hubbard ME, Lockyer J, Podolak O, Dammavalam VM, Grady M, Nance M, Scheiman M, Samadani U, Master CL. Eye Tracking as a Biomarker for Concussion in Children. Clin J Sport Med. 2020 Sep;30(5):433-443. doi: 10.1097/JSM.0000000000000639. PMID 30095503
- [Background] Ciuffreda KJ, Joshi NR, Truong JQ. Understanding the effects of mild traumatic brain injury on the pupillary light reflex. Concussion. 2017 Aug 3;2(3):CNC36. doi: 10.2217/cnc-2016-0029. eCollection 2017 Nov. PMID 30202579
- [Background] Thiagarajan P, Ciuffreda KJ. Pupillary responses to light in chronic non-blast-induced mTBI. Brain Inj. 2015;29(12):1420-5. doi: 10.3109/02699052.2015.1045029. Epub 2015 Jul 16. PMID 26182230
- [Background] Walsh DV, Capo-Aponte JE, Beltran T, Cole WR, Ballard A, Dumayas JY. Assessment of the King-Devick(R) (KD) test for screening acute mTBI/concussion in warfighters. J Neurol Sci. 2016 Nov 15;370:305-309. doi: 10.1016/j.jns.2016.09.014. Epub 2016 Sep 11. PMID 27646958
- [Background] Anderson M, Elmer J, Shutter L, Puccio A, Alexander S. Integrating Quantitative Pupillometry Into Regular Care in a Neurotrauma Intensive Care Unit. J Neurosci Nurs. 2018 Feb;50(1):30-36. doi: 10.1097/JNN.0000000000000333. PMID 29303836
- [Background] Chen JW, Gombart ZJ, Rogers S, Gardiner SK, Cecil S, Bullock RM. Pupillary reactivity as an early indicator of increased intracranial pressure: The introduction of the Neurological Pupil index. Surg Neurol Int. 2011;2:82. doi: 10.4103/2152-7806.82248. Epub 2011 Jun 21. PMID 21748035
- [Background] McNett M, Moran C, Janki C, Gianakis A. Correlations Between Hourly Pupillometer Readings and Intracranial Pressure Values. J Neurosci Nurs. 2017 Aug;49(4):229-234. doi: 10.1097/JNN.0000000000000290. PMID 28661946
- [Background] Voelker R. Eye-Tracking Test Approved to Help Diagnose Concussion. JAMA. 2019 Feb 19;321(7):638. doi: 10.1001/jama.2019.0509. No abstract available. PMID 30778585
- [Background] Covassin T, Elbin RJ 3rd, Stiller-Ostrowski JL, Kontos AP. Immediate post-concussion assessment and cognitive testing (ImPACT) practices of sports medicine professionals. J Athl Train. 2009 Nov-Dec;44(6):639-44. doi: 10.4085/1062-6050-44.6.639. PMID 19911091
- [Background] Iverson GL, Schatz P. Brief iPad-Based Assessment of Cognitive Functioning with ImPACT(R) Pediatric. Dev Neuropsychol. 2019 Jan-Feb;44(1):43-49. doi: 10.1080/87565641.2018.1545844. Epub 2018 Nov 22. PMID 30466316
- [Background] Howell DR, Osternig LR, Chou LS. Detection of Acute and Long-Term Effects of Concussion: Dual-Task Gait Balance Control Versus Computerized Neurocognitive Test. Arch Phys Med Rehabil. 2018 Jul;99(7):1318-1324. doi: 10.1016/j.apmr.2018.01.025. Epub 2018 Feb 16. PMID 29457997
- [Background] Bell DR, Guskiewicz KM, Clark MA, Padua DA. Systematic review of the balance error scoring system. Sports Health. 2011 May;3(3):287-95. doi: 10.1177/1941738111403122. PMID 23016020
- [Background] Capó-Aponte, JE, Urosevich TG, Walsh DV, Temme LA, & Tarbett AK. Pupillary light reflex as an objective biomarker for early identification of blast-induced mTBI. Journal of Spine S4:004, 2013.
- [Background] Coronado VG, McGuire LC, Sarmiento K, Bell J, Lionbarger MR, Jones CD, Geller AI, Khoury N, Xu L. Trends in Traumatic Brain Injury in the U.S. and the public health response: 1995-2009. J Safety Res. 2012 Sep;43(4):299-307. doi: 10.1016/j.jsr.2012.08.011. Epub 2012 Aug 25. PMID 23127680